CLINICAL TRIAL: NCT01455844
Title: A Randomized, Placebo-controlled, Double-blind, Dose-ranging, Multi-centered Trial to Evaluate the Safety and Efficacy of NKPL66 (CaPre™) in the Treatment of Mild-to-high Hypertriglyceridemia
Brief Title: TRIal For Efficacy of Capre on hyperTriglyceridemiA
Acronym: TRIFECTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grace Therapeutics Inc. (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRT-API-NKPL66-CT-PII
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Hypertriglyceridemia
Keywords: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CaPre 1.0g (Experimental)
  Interventions: Drug: CaPre (TM)
- CaPre 2.0g (Experimental)
  Interventions: Drug: CaPre (TM)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CaPre (TM) — CaPre™ 1.0g + Placebo 1.0g daily for 12 weeks.
  Arms: CaPre 1.0g
Other: Placebo — 2.0g Placebo (Microcrystalline cellulose) daily for 12 weeks
  Arms: Placebo
Drug: CaPre (TM) — CaPre™ 2.0g daily for 12 weeks
  Arms: CaPre 2.0g

SUMMARY:
The purpose of this study is to determine whether CaPre(TM), given at doses 1.0g or 2.0g for 12 weeks, has an effect on fasting plasma triglycerides in patients with mild to high hypertriglyceridemia as compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18 to 75 years.
* Fasting plasma levels of TG ≥ 2.28 and <10 mmol/L (200 and 877 mg/dL) on two occasions within 2 weeks (screening and pre-randomization visits).
* Patients who are currently not on pharmacotherapy for hyperlipidemia and according to the judgement of the physician and Canadian Guidelines for the Diagnosis and Treatment of Dyslipidemia initiation of drug therapy is not indicated for the duration of the study.
* Patients currently treated with statins and according to the judgement of the physician and the Canadian Guidelines for the Diagnosis and Treatment of Dyslipidemia a change in their current drug regimen is not indicated for the duration of the study.
* Patients treated with statin must be on stable dose for at least 6 weeks prior to screening.
* Patients are willing follow the NCEP Step 1 Diet (see Appendix 4) for the duration of the study.
* Female participants of childbearing potential (i.e. not surgically sterilized or post-menopausal greater than one year) must have negative serum pregnancy test and must be using an effective birth control method, defined as:

  1. continuous use of oral or long acting injected contraceptive for at least 2 months prior to study entry, or;
  2. use of an intra-uterine device or implantable contraceptive, or;
  3. use of double barrier methods of birth control
* Patients are at least 80% compliant with the study medication during the placebo lead in phase.

Exclusion Criteria:

* Any concomitant medication which in the opinion of the investigator would preclude the patient from successfully participating in the study.
* Women who are pregnant or that are breast feeding.
* Participation in another clinical trial within 30 days from initiation of the study.
* Participants with a high risk for cardiovascular disease; (The definition of high-risk individuals will follow that of the 2009 Canadian Guidelines and include a) FRS >= 20% 10-year risk; b) All patients with uncontrolled diabetes (DCA guidelines) and c) Evidence of atherosclerosis -when this evidence was ascertained when clinically indicated);
* Systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg. In diabetic patients, systolic blood pressure > 130 mmHg and/or diastolic blood pressure > 90 mmHg.
* History of stroke, intermittent claudication or transient ischemic attack.
* Known unstable (uncontrolled) cardiac disease , within the last 6 months.
* Patient with a clinically significant abnormal ECG at screening.
* Patients with uncontrolled diabetes mellitus, with HbA1c > 7.0%.
* Known diagnosis of hypoglycemia.
* Evidence of active renal disease indicated by a fasting estimated glomerular filtration rate (eGFR) of < 60 ml/min per 1.73 m2.
* Increased plasma levels (>ULN) of amylase (as per respective lab upper limits) and / or lipase (>160 IU/L) or any indication of pancreatitis pancreatitis (increased alcohol consumption, gallstones).
* History of pancreatitis.
* Use of any lipid lowering medication other than statins or ezetimibe(e.g niacin, fibrates) and/or lipid lowering NHP within 6 weeks prior to the screening visit.
* Intake of > 2 servings per week of fish or regimented use of fish oil/omega-3 supplements within 6 weeks prior to the screening visit.
* Known HIV or Hepatitis B or C positive.
* Patients with uncontrolled asthma as defined by the 2010 Consensus Summary of the Canadian Thoracic Society.
* Known seafood allergy or allergy to any of the medicinal or non-medicinal ingredients of the study medication and placebo, including:

  1. Omega-3 fatty acids (including EPA and DHA)
  2. Phospholipids (mainly phosphatidylcholine)
  3. Astaxanthin
  4. Microcrystalline cellulose
* Coagulopathy or on anticoagulants. Platelet aggregation inhibitors (such as aspirin or clopidogrel but not heparin) are permitted in the study; patients taking both aspirin and clopidogrel are not permitted in the study.
* Unable or unwilling to comply with the protocol.
* Patient reported weight was not stable for the past 6 months (within 3kg variation).
* Consumption of more than 14 standard alcoholic drinks a week.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percent (%) change in triglycerides between the baseline and the 12-week assessment visit. | 12 weeks

SECONDARY OUTCOMES:
Absolute change in triglycerides between the baseline and the 12-week assessment visit. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Genest, MD, FRCP(C), Principal Investigator — Cardiology Division, MUHC
Locations (38):
- Canada (38):
  - Cardiology Research, Edmonton, Alberta
  - Kelowna, British Columbia
  - Medical Arts Health Research Group, Penticton, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - CookMed Research, Victoria, British Columbia
  - First Line Medical Services Ltd, St. John's, Newfoundland and Labrador
  - White Hills Medical Clinic, St. John's, Newfoundland and Labrador
  - Scisco Clinical Research, Cornwall, Ontario
  - Corunna Medical Resarch Centre, Corunna, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - MD-Medical Professional Corporation, Hamilton, Ontario
  - Source Unique Research Inc., Hawkesbury, Ontario
  - Bagot Street Medical Centre, Kingston, Ontario
  - KGK Synergize Inc., London, Ontario
  - Milestone Research, London, Ontario
  - Robarts Research Institute, London, Ontario
  - SPARC, Siebens-Drake Research Institute, London, Ontario
  - S & G Clinical Research, Mississauga, Ontario
  - SKDA Research Inc., Newmarket, Ontario
  - Niagara Falls, Ontario
  - Centre Medical Phoenix, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - Canadian Phase Onward, Toronto, Ontario
  - Source Unique Research Inc., Dollard-des-Ormeaux, Quebec
  - CLIN DE MED Grand-Mere, Grand-Mère, Quebec
  - Diex Research Montreal Inc., Montreal, Quebec
  - Institut de recherches cliniques de Montréal (IRCM), Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Dynamik Research Inc., Pointe-Claire, Quebec
  - Kells Medical Research, Pointe-Claire, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc, Québec, Quebec
  - Clinique Médicale St-Louis, Québec, Quebec
  - Pro-Recherche Inc., Saint Romuald, Quebec
  - Centre médical-des-carrières, Saint-Marc-des-Carrieres, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec